CLINICAL TRIAL: NCT03173716
Title: (RTMPE in the ICU) The Impact of Real-Time Myocardial Perfusion Echocardiography on Diagnostic Confidence and Subsequent Management of Myocardial Ischemia in the Intensive Care Unit
Brief Title: Real-Time Myocardial Perfusion Echocardiography in the ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Patricia A. Pellikka, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-009331
Record Dates: First submitted 2017-05-23; First posted 2017-06-02 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Perfusion Imaging
Keywords: DEFINITY contrast
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): DEFINITY contrast will be prepared according to package insert instructions. A dose of 1.5 mL activated DEFINITY diluted in 28.5 of preservative free saline to constitute a total volume of 30 mL will be infused at a rate of 90-120 mL/hr (1.5-2.0 mL/min). RTMPE will be performed.
  Interventions: Procedure: Definity
- Control Arm (No Intervention): Echocardiograms will be performed without the use of DEFINITY contrast/RTMPE.

INTERVENTIONS:
Procedure: Definity — Real-Time Myocardial Perfusion Echocardiography (RTMPE) will be performed as opposed to the standard echocardiogram (TTE) of the control arm
  Arms: Intervention Group

SUMMARY:
This study is being done to find out if and how much the use of RTMPE improves a provider's confidence in the diagnosis they assign. This is important because the use of RTMPE may decrease the need for any additional invasive testing.

DETAILED DESCRIPTION:
The finding of elevated troponins and regional wall motion abnormalities on echocardiography in the absence of other signs of acute coronary syndrome among the intensive care population creates a diagnostic challenge for evaluation. Sometimes these ill patients undergo invasive coronary angiography to rule out acute thrombosis. Real-Time Myocardial Perfusion Echocardiography (RTMPE) is a safe and accurate imaging modality to assess perfusion and can be performed in the resting state at the bedside in the intensive care unit (ICU) to help stratify the likelihood intracoronary thrombosis as the etiology for abnormal troponins and/or echocardiography. The primary aim of this study is to evaluate the impact of RTMPE on providers' diagnostic confidence using a 5-point Likert scale for patients that receive a standard transthoracic echocardiogram (TTE) compared to patients that receive RTMPE. The RTMPE to assess perfusion will be added to the standard transthoracic echocardiogram in approximately 24 patients undergoing evaluation of myocardial ischemia in medical or surgical ICUs. The caring provider will complete a web-based survey regarding their confidence in the diagnosis prior to and after the study in both groups. The images will be interpreted by an experienced cardiologist and results will be made available in the medical record. The difference in diagnostic confidence scores will be analyzed using the Wilcoxon signed-rank test. The secondary aims are to assess the management and outcomes in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age ≥ 18 years
2. Located in a designated ICU
3. TTE ordered by the primary care team
4. Significant delta in troponin trend
5. Concern for myocardial ischemia
6. Women of child-bearing potential must have a clinical negative pregnancy test result
7. Experienced sonographer available to complete RTMPE portion of the exam
8. Provider willing to complete the study survey

Exclusion Criteria:

1. Adults < 18 years
2. Contraindication to echo contrast administration
3. Location other than an ICU
4. No significant delta in troponin trend

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Diagnostic Confidence Post-Echocardiography | through study completion, anticipated 1 year
  5-point Likert scale will be used to assess providers' diagnostic confidence

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Pellikka, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials